CLINICAL TRIAL: NCT00497848
Title: Individual Versus System Orientated Interventions in Handling Drug Related Problems in People With Schizophrenia
Brief Title: The Compliance Project Concerning People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of the Interior and Health, Denmark (Other Government)
Responsible Party: MD, PhD Bent Nielsen, Department of Psychiatry, Odense, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: MIH, Denmark
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2007-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- motivational interviewing (Active Comparator)
  Interventions: Behavioral: motivational interviewing
- The System Orientated Intervention (Experimental)
  Interventions: Other: The System-Orientated Intervention

INTERVENTIONS:
Behavioral: motivational interviewing — An individual intervention building on the "Motivational Interviewing" by Miller and Rollnick. Several studies has proved effectiveness of this therapy form in improving drug compliance. Patients will be offered individual motivational therapy
  Other Names: compliance therapy
  Arms: motivational interviewing
Other: The System-Orientated Intervention — Principles in this intervention come from "Clinical Risk Managing" and quality assurance. It focuses on daily problems in drug handling, including dropping out of drug therapy, by looking at the system as a whole.Some cases, where patients dropped out of drug therapy will be carefully analysed in order to identify week points in the system, and subsequently alter the instructions for drug therapy, information, reminders and so on.
  Other Names: Clinical Risk Managing in Handling Compliance Problems
  Arms: The System Orientated Intervention

SUMMARY:
The purpose of this study is to determine whether individual and/ or system orientated interventions can help the problem of people with schizophrenia dropping out of their drug treatment

DETAILED DESCRIPTION:
50% of people with schizophrenia do not take the prescribed medication leading to repeating relapses with loss of social and cognitive skills.

The individual intervention is based on "Motivational Interviewing" by Miller and "Concordance Strategies" by R. Gray.It is a cognitive behavioral therapy.

The system orientated intervention is building on principles from quality assurance and clinical risk managing. It seeks to improve the quality in the medical treatment by use of standards, monitoring, audit and root cause analysis,and thereby trying to find weak points in the system and subsequently improve the common practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of schizophrenia or schizoaffective psychosis
* 23 years or more
* Ethnic dane
* Living in the city of Odense.

Exclusion Criteria:

* not subject to legal action

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
compliance assessed on a compliance-scale | follow-up time 6 months

SECONDARY OUTCOMES:
assessment on a variety of scales concerning subjective well-being, GAF, PANSS-remission,CGI, side-effects. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bent Nielsen, Ph. D., Study Director — University of Southern Denmark
Locations (1):
- Department of psychiatry, Odense University Hospital, Odense, Denmark